CLINICAL TRIAL: NCT07289035
Title: Exploratory Study to Evaluate the Safety and Tolerability of Tamoxifen Citrate in the Treatment of Cystic Fibrosis in Patients Without Mutations Currently Eligible for Therapy With CFTR Modulator Drugs
Brief Title: Early Study on Tamoxifen Safety/Tolerability in Cystic Fibrosis Patients Unable to Use CFTR Modulators.
Acronym: TMX
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRCFC-TAMOXI063; 2024-519657-11-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-20; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-08

CONDITIONS: Cystic Fibrosis - Complete
Keywords: Cystic Fibrosis; Tamoxifen; CaCC
MeSH Terms: conditions — Cystic Fibrosis | interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tamoxifen citrate (Experimental): Patients will receive TMX 20 mg/day, in the morning. The choice of this dosage is based on pharmacokinetic and pharmacodynamic data in the literature in patients with breast cancer. Based on this scientific evidence, the dose of 20 mg/day is the minimum dose to ensure safety and efficacy of treatment.
  Women should start treatment with TMX between 8 and 12 days after the onset of menstruation. A longer screening period to allow for this timing will not be considered a protocol violation. Men will start treatment at V2 (day 1) and continue at home for 24 weeks. After screening, visits will be performed on the first day of TMX administration (baseline) and after 4, 8, 12, 16, and 24 weeks. Patients will discontinue TMX treatment at week 24 and will be followed for an additional 4 weeks for safety evaluation.
  Interventions: Drug: Tamoxifen Citrate 20Mg Tab

INTERVENTIONS:
Drug: Tamoxifen Citrate 20Mg Tab — One tablet per day (20 mg/day), in the morning.
  Other Names: TMX

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of TMX in adults patients with cystic fibrosis who do not have mutations currently eligible for therapy with modulator drugs.

The main questions it aims to answer is:

. What medical problems do participants have when taking drug TMX?

Participants will:

* Take drug TMX every day for 6 months
* Visit the clinic once every 28 days for checkups and tests

DETAILED DESCRIPTION:
Normal airways regulate the volume of airway surface liquid (ASL) through the activation of both cyclic adenosine monophosphate (cAMP) and Ca2+-dependent ion channels. In cystic fibrosis, the genetic defect causes a deficiency of cAMP-dependent CFTR (Cystic Fibrosis Transmembrane Conductance Regulator) activity, leading to reduced Cl- and water secretion from airway epithelial cells and the consequent accumulation of mucus, facilitating bacterial and fungal infections. Women with CF have reduced survival compared with men with CF, although the mechanisms underlying this sex-related disadvantage are unknown. Despite the lack of CFTR, CF airways maintain a limited ability to regulate ASL volume, as ATP release, induced by breathing, activates purinergic pathways that increase intracellular Ca2+ concentration to stimulate an alternative Cl- secretion pathway. It has been hypothesized that estrogen might influence this pathway by reducing the ability of airway epithelia to adequately respond to nucleotides. They found that UTP-mediated Cl- secretion was reduced during periovulatory estrogen peaks in both CF and healthy women. Estrogen also inhibited Ca2+ signaling and ASL volume homeostasis in both non-CF and CF airway epithelia by attenuating Ca2+ influx. 17ß-estradiol inhibits the intracellular Ca2+ signaling, thus impairing the activity of calcium-activated chloride channels (CaCC). This suggests that antiestrogens, such as tamoxifen, could be beneficial in the treatment of CF lung diseases because they may increase Cl- secretion in the airways.

It has been demonstrated that TMX can restore CaCC function by inhibiting estrogen signaling. Furthermore, authors showed that TMX can directly activate CaCC regardless of estrogen signaling, therefore generating a significant amount of chloride current.

The results of these experiments indicate that:

* TMX can increase CaCC currents through two mechanisms:

  * Indirectly, as an antagonist of the negative effect of 17β-estradiol on the currents
  * Directly, regardless of the antiestrogen effect, by acting on CaCC, the alternative chloride transport pathway
* The action of TMX is not affected by the different class of CFTR mutations since it regulates CaCC
* The effect of TMX on CaCC currents is long-lasting and quantitatively significant, superior to the CFTR-dependent currents obtained from the combination of ivacaftor and lumacaftor
* Both women and men can benefit from TMX
* TMX antagonizes the inhibitory action of estradiol E2 on CaCC currents: TMX could counteract the negative effects of estrogens on CaCC currents during the periovulatory period (about 1 week per month) and acts directly on CaCC currents during all remaining days
* It can be used in combination with other therapeutic agents: given the complexity of intracellular trafficking and the short half-life of mutant CFTR proteins, it is conceivable that the currently available CFTR modulators will improve but not cure cystic fibrosis. Therefore, the treatment of cystic fibrosis may require the combination of different therapeutic agents. TMX treatment could be complementary and synergistic with CFTR modulators.

In conclusion, although effective therapies for CF have been already authorized in the European Union, the use of tamoxifen citrate is justified by the current scientific literature and preclinical data. Patients with CF should benefit from this treatment. Importantly, given its mechanism of action, TMX is expected to be beneficial for patients both with F508del CFTR mutation and other rare variants that still remain orphan of therapies. It follows that the European Commission has considered TMX treatment as a possible clinically relevant advantage for patients with CF.

Based on the results emerged from different studies, the European Commission has granted orphan designation (EU/3/17/1877) to GB Pharma S.r.l. for tamoxifen citrate for the treatment of cystic fibrosis.

Primary Objective The study aims to evaluate the safety and tolerability of TMX in patients with cystic fibrosis who do not have mutations currently eligible for therapy with modulator drugs.

Secondary Objectives

The study also aims to evaluate the effects of TMX on:

* lung function
* quality of life
* pulmonary exacerbations
* hospitalizations for pulmonary exacerbations
* antibiotic cycles
* BMI
* sputum microbiology
* sweat test

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if they meet all the following inclusion criteria at Visit 1:

1. Subjects of both sexes, affected by cystic fibrosis, attending the CF Center in Verona
2. Patients who do not have mutations currently eligible for therapy with CFTR modulator drugs
3. Age 18 years or older
4. Predicted forced expiratory volume in 1 second (ppFEV1) ≥ 40% and ≤ 90% (of the predicted value for people of their age, sex, and height) before bronchodilator administration
5. Stable routine CF therapy in terms of dose and medication (inhaled antibiotic cycles, bronchodilator, anti-inflammatory, inhaled corticosteroid, physiotherapy technique/schedule) within 28 days prior to Day 1
6. Clinically stable respiratory disease within 3 weeks before Day 1 (first dose of study drug)
7. Subjects able to perform reliable and reproducible pulmonary function test maneuvers
8. Subjects able to communicate well with the investigator, understand, and comply with the study requirements
9. Female subjects must have a negative serum pregnancy test
10. Sexually active subjects able to follow the contraceptive methods defined within the protocol (non-hormonal contraception) during the study and for 2 months after study discontinuation
11. Signed informed consent for participation in the study and for the processing of personal data.

Exclusion Criteria:

Patients will be excluded if one or more of the following criteria are met at Visit 1:

1. Patients on any CFTR modulator therapy
2. Pulmonary exacerbations within 3 weeks before Day 1 (first dose of study drug)
3. Changes in therapy for lung disease within 3 weeks before Day 1 (first dose of study drug)
4. Family and/or personal history of thromboembolism and thromboembolic conditions up to 1st-degree relatives
5. Documented hereditary thrombophilia (hypercoagulability), e.g., protein C, protein S, and antithrombin deficiency; factor V G169A Leiden, prothrombin G20210A (PT20210A), elevated factor VIII levels, hereditary dysfibrinogenemia
6. History of solid organ or hematopoietic transplant
7. History of hypersensitivity to the study drug or drugs of similar chemical classes or any excipients
8. History or presence of prolonged QT interval (QTcB > 450 msec)
9. History of malignancy in any organ system (other than localized basal cell carcinoma of the skin) in the last 5 years
10. Hemoglobin levels < 9.0 g/dl
11. Any surgical or medical condition that may significantly alter the absorption, distribution, metabolism, or excretion of drugs, or that may jeopardize the subject in case of participation in the study
12. History of immunodeficiency diseases
13. History of drug or alcohol abuse
14. History of any disease or condition that, in the investigator's opinion, could confound the study results
15. Abnormal liver function, defined as ≥ 3 times the upper limit of normal (ULN) for any of the following: serum aspartate transaminase (AST), serum alanine transaminase (ALT), total bilirubin.
16. Presence at baseline visit of endometrial polyps or vaginal symptoms (e.g., blood discharge, spotting, staining)
17. Participation in a clinical study where an investigational drug was administered within 30 days prior to enrollment in the study or 5 half-lives of the study drug, whichever is longer
18. Female patients who are pregnant or breastfeeding or who wish to become pregnant during the clinical study period and within one month after the end of the study
19. Female patients of childbearing potential who do not use adequate contraception. A woman is considered of childbearing potential (WOCBP), i.e., fertile, after menarche and until reaching post-menopause, unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. A postmenopausal state is defined as the absence of menstruation for 12 months without an alternative medical cause. An elevated follicle-stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormone replacement therapy. However, in the absence of 12 months of menstrual cycle, a single FSH measurement is not sufficient.* *Low failure rate contraceptive methods (less than 1% per year) if used consistently, including: some intrauterine devices, abstinence, or vasectomized partner. Contraception must be maintained until 1 month after the last visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Calculating between baseline and week 24
  The primary endpoint of this study will be evaluated by calculating between baseline and week 24 the incidence of serious adverse events (SAEs), treatment-emergent adverse events (TEAEs) and treatment discontinuation due to AEs. In addition, frequency of specific, indication-relevant adverse events (e.g., thromboembolic events, elevation of liver enzymes, pulmonary exacerbations) and cumulative AE analyses, such as the number of AEs per patient, will be also evaluated.

SECONDARY OUTCOMES:
Changes in respiratory function values | From baseline to week 24
  The relative change from baseline to week 24 in ppFEV1
Changes in pulmonary exacerbation | Up to week 24
  The number of pulmonary exacerbations up to week 24 and the time to the first pulmonary exacerbation up to week 24
Changes in hospitalizations | From baseline to week 24
  The number of hospitalizations for cystic fibrosis lasting > 24 hours and the time to the first hospitalization for cystic fibrosis
Changes in quality of life | From baseline to week 24
  The absolute change in the respiratory domain score of the Cystic Fibrosis Questionnaire-Revised (CFQ-R) (the more the value increases, the greater the perceived well-being)
Changes in antibiotic use | Up to week 24
  * the use of intravenous antibiotics during the study (total number of days of intravenous antibiotics for sino-pulmonary signs and symptoms up to week 24)
  * the use of oral antibiotics during the study (total number of days of oral antibiotics for sino-pulmonary signs and symptoms up to week 24)
Changes in BMI | From baseline to week 24
  Changes in BMI from baseline to week 24
Changes in sputum microbiology | From screening to week 24
  Changes in sputum microbiology from screening to week 24
Sweat test - Changes in amount of chloride | At the beginning and end of the study
  Changes in the amount of chloride measured with the sweat test

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Fibrosi Cistica - AOUI Verona, Verona, Veneto, Italy

IPD SHARING:
Plan to Share IPD: No